CLINICAL TRIAL: NCT05649631
Title: The Effect of Low Sodium Diet on Idiopathic Hyperaldosteronism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, Director,head of Endocrinololgy,Principal Investigator,Clinical Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ruijin-2020-294
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Primary Aldosteronism Due to Adrenal Hyperplasia (Bilateral)
MeSH Terms: interventions — Sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal sodium diet(100mmol/d) (Experimental)
  Interventions: Dietary Supplement: Sodium
- Low sodium diet(50mmol/d) (Experimental)
  Interventions: Dietary Supplement: Sodium

INTERVENTIONS:
Dietary Supplement: Sodium — 50 IHA patients were randomized into two groups with low sodium (50mmol/d) and normal sodium (100mmol/d) without potassium supplement. A 14 days dietary intervention was performed respectively to compare the changes in blood pressure (BP) and serum potassium in two groups.

SUMMARY:
This study was a single-center randomized controlled trial which lasted 14 days and consisted of two stages (run-in period (stage I) and intervention period (stage II) each contain 7 days without potassium supplement. If participants meet the enrollment criteria at the end of stage I, they were assigned to the low sodium group (50mmol/d) or normal sodium group (100mmol/d), and then continued to finish stage II. The primary outcome was the change in serum potassium after exposure to normal sodium / low sodium diet and the secondary outcome was the assessment of BP change following a normal sodium / low sodium diet. Patients were given nifedipine controlled-release tablets 30 mg/d to lower blood pressure and were not provided any potassium supplements during the two stages. If the subject has an increase in BP (>180/110 mmHg), the dose of nifedipine controlled-release tablets will be increased to 60 mg/d. Patients will be withdrawn from the study if they cannot tolerate the diet or their serum potassium were below 2.8 mmol/L.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years;
2. diagnosed as PA by SIT;
3. no lateralization of aldosterone secretion during AVS;
4. serum potassium ≥ 2.8 mmol/L after the stage I.

Exclusion Criteria:

1. Impaired renal function (Ccr<60 ml/min);
2. Impaired liver function (ALT, AST > 2.5 times upper limit of normal);
3. Patients with heart failure (NYHA≥ class 3 or EF < 50%);
4. Patients with stroke or acute infarction in the last 6 months;
5. Patients who are pregnant or breastfeeding;
6. Patients who cannot tolerate dietary arrangements;
7. Patients with history of malignant tumors in the last 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the change in serum potassium after exposure to normal sodium / low sodium diet | 2 weeks

SECONDARY OUTCOMES:
The secondary outcome was the assessment of BP change following a normal sodium / low sodium diet. | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yiran Jiang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou L, Jiang Y, Zhang C, Su T, Jiang L, Zhou W, Zhong X, Wu L, Wang W. Effects of a low-sodium diet in patients with idiopathic hyperaldosteronism: a randomized controlled trial. Front Endocrinol (Lausanne). 2023 Apr 19;14:1124479. doi: 10.3389/fendo.2023.1124479. eCollection 2023. PMID 37152926